CLINICAL TRIAL: NCT03808064
Title: Community-based Intervention for Cervical Cancer Screening Uptake in a Semi-urban Area of Pokhara Metropolitan, Nepal: A Cluster Randomized Controlled Trial (COBIN-C)
Brief Title: Community-based Intervention for Cervical Cancer Screening Uptake in Nepal
Acronym: COBIN-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Aamod Dhoj Shrestha, PhD Fellow, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ADS18
Record Dates: First submitted 2019-01-10; First posted 2019-01-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Cervical Cancer Screening
Keywords: Cervical cancer screening; Community health worker; Community-based; Female community health volunteers; Non-communicable diseases; Randomized controlled trial; Nepal
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): After randomization, the FCHVs in the intervention arm will receive training, health education materials and a recording register. After receiving training, they will educate women of their respective ward on cervical cancer screening and prevention through home visits and maintain records in their service register.
  Interventions: Behavioral: FCHV home visit
- Control arm (No Intervention): There won't be any intervention in the control arm.

INTERVENTIONS:
Behavioral: FCHV home visit — Behavioral: FCHV visit Female Community Health Volunteer will visit selected households 3 times a year for providing health promotion messages Other Name: FCHV Home Visit
  Arms: Intervention arm

SUMMARY:
This study aims to evaluate the effect of a Female Community Health Volunteer (FCHV) led community-based educational intervention through home visits increasing cervical cancer screening uptake.

DETAILED DESCRIPTION:
Cervical cancer is the major cause of cancer deaths among women in Nepal. Screening is one of the most effective tools for early diagnosis, prevention, and treatment. However, skilled health professionals and tools available for cervical cancer screening are limited in low and middle-income countries (LMICs) including Nepal. The World Health Organization (WHO) and Alliance for Cervical Cancer Prevention (ACCP) recommends that countries, areas, or institutions seeking to initiate or strengthen cervical cancer screening programs should consider introducing or expanding Visual Inspection with Acetic acid (VIA) until more appropriate and affordable HPV-based tests become available. 'National Guideline for Cervical Cancer Screening and Prevention in Nepal, 2010' includes VIA as a screening method for cervical cancer. Current studies reveal Nepalese women's participation in cervical cancer screening is low. Thus, there is a need for appropriate, cost-effective and sustainable interventions to increase VIA screening uptake at the primary health care level across Nepal.

The primary objective of this study is to evaluate the effect of a Female Community Health Volunteer (FCHV) led community-based educational intervention through home visits increasing cervical cancer screening uptake. The primary outcome of the study is to increase the cervical cancer-screening uptake in the intervention group. This will be the first community-based cluster-randomized trial designed to mobilize FCHVs for increasing cervical cancer screening uptake in Nepal.

ELIGIBILITY:
Inclusion Criteria:

* All women of age group 30-60 years who were recruited in the COBIN Wave I survey

Exclusion Criteria:

* Women who are not able to give consent
* Severely ill,
* Pregnant or less than 6 weeks after delivery,
* Who is already diagnosed with cervical pre-cancer and cancer
* With a history of total hysterectomy
* Who are reluctant to participate in the study or unable to complete the interview

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 690 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2020-12-26 (Actual); Study Completion 2020-12-26 (Actual)

PRIMARY OUTCOMES:
The increase in the number of participants attending cervical cancer screening after education intervention | One year
  The effect of Female Community Health Volunteers led community based educational intervention through home visits for increasing cervical cancer screening uptake will be evaluated by comparing the baseline with follow up study.

CONTACTS AND LOCATIONS:
Overall Officials: Aamod D Shrestha, MPH, Principal Investigator — Department of Public Health, Aarhus University, Aarhus, Denmark
Locations (1):
- Nepal Development Society, Pokhara, Gandaki, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dhoj Shrestha A, Gyawali B, Shrestha A, Shrestha S, Neupane D, Ghimire S, Campbell C, Kallestrup P. Effect of a female community health volunteer-delivered intervention to increase cervical cancer screening uptake in Nepal: a cluster randomized controlled trial. Prev Med Rep. 2022 Aug 12;29:101948. doi: 10.1016/j.pmedr.2022.101948. eCollection 2022 Oct. PMID 36161136
- [Derived] Shrestha AD, Neupane D, Ghimire S, Campbell C, Kallestrup P. Community-based intervention for cervical cancer screening uptake in a semi-urban area of Pokhara Metropolitan, Nepal (COBIN-C): study protocol for a cluster-randomized controlled trial. Trials. 2021 Jan 26;22(1):94. doi: 10.1186/s13063-021-05049-3. PMID 33499911